CLINICAL TRIAL: NCT05522465
Title: Short-course High-dose Prednisone and Dexamethasone in Children With Immune A Multicenter, Randomized Controlled Study of Thrombocytopenia
Brief Title: Short-course High-dose Prednisone and Dexamethasone in Children With ITP
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fujian Medical University Union Hospital (Other)
Collaborators: The First Affiliated Hospital of Xiamen University (Other); Zhangzhou Affiliated Hospital of Fujian Medical University (Other); Quanzhou First Hospital (Other); Nanping First Hospital Affiliated to Fujian Medical University (Unknown); The Second Hospital of Anhui Medical University (Other); The Affiliated Hospital Of Guizhou Medical University (Other); Longyan City First Hospital (Other); The Affiliated Hospital of Putian University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022YF025-01
Record Dates: First submitted 2022-08-29; First posted 2022-08-31 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-02

CONDITIONS: Immune Thrombocytopenia; Glucocorticoids; Child, Only
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Prednisone; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- prednisone group (Experimental): prednisone 4mg/kg.d
  Interventions: Drug: Prednisone
- Dexamethasone (Active Comparator): Dexamethasone 0.6mg/kg.d
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Prednisone — Prednisone 4mg/kg.d, d1-4
  Arms: prednisone group
Drug: Dexamethasone — Dexamethasone 0.6mg/kg.d, d1-4
  Arms: Dexamethasone

SUMMARY:
Comparison of the efficacy and safety of short-course high-dose prednisone and dexamethasone in the treatment of children with newly diagnosed immune thrombocytopenia (ITP)

ELIGIBILITY:
Inclusion Criteria:Subjects enrolled in this study must meet all of the following criteria:

1. Meet the ITP diagnostic criteria, within 3 months of the first diagnosis
2. Age > 28 days and ≤ 14 years old
3. Untreated PLT<20×109/L, or PLT<30×109/L after 1 week of intravenous gamma globulin (IVIG) treatment
4. Have signed the informed consent

Exclusion Criteria:Anyone who has any of the following conditions will not enter the clinical study:

1. Intracranial hemorrhage or severe gastrointestinal or urinary tract hemorrhage requiring emergency treatment, such as simultaneous use of platelet transfusion and thrombopoietic drugs (recombinant human thrombopoietin, eltrombopag, etc.)
2. Received glucocorticoid therapy within 6 months
3. Menstrual female children
4. Patients with underlying diseases such as tumor diseases, autoimmune diseases or genetic diseases
5. Patients who have received radiotherapy and chemotherapy
6. There are contraindications to the use of glucocorticoids (hypertension, glaucoma, peptic ulcer, etc.)
7. There are any significant abnormal coexisting diseases or mental illnesses that affect the patient's life safety and compliance, and affect informed consent, research participation, follow-up or interpretation of results

Ages: 29 Days to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 608 (Estimated)
Dates: Start 2022-10-11 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
initial treatment response | 30 days after treatment
  Platelet count after glucocorticoid therapy 1 month

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 1 month
  Incidence of Treatment-Emergent Adverse Events occurring within 1 month of glucocorticoid therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Children with newly dignosed ITP, Fujian, Fujian, China